CLINICAL TRIAL: NCT05448274
Title: An Intervention Study to Explore Potential Metabolic Effects of Ruminococcus Torques Strain ATCC 27756 in Healthy Adults
Brief Title: The Effects of a Ruminococcus Torques Strain Bacterium in Healthy Adults.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oluf Pedersen (Other)
Collaborators: University of Copenhagen (Other); Technical University of Denmark (Other); University Hospital, Gentofte, Copenhagen (Other)
Responsible Party: Sponsor-Investigator, Oluf Pedersen, Professor, MD, University Hospital, Gentofte, Copenhagen
Organization: University Hospital, Gentofte, Copenhagen (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: H-21075670
Record Dates: First submitted 2022-06-28; First posted 2022-07-07 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Overweight; Healthy
Keywords: Metabolism; Microbiota; Ruminococcus torques
MeSH Terms: conditions — Overweight

STUDY DESIGN:
Intervention Model Description: A crossover study where subjects recieve placebo or Ruminococcus torques on two different study days with three to six weeks of wash-out between the study days.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blinded study where both the investigator (the physician), care provider (nurse) and the participants are blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): The placebo will consist of solely glycerol-phosphate-buffered isotonic saline.
  Interventions: Biological: Placebo
- Ruminococcus torques (Experimental): 10^11 live bacterial cells in glycerol-phosphate-buffered isotonic saline
  Interventions: Biological: Ruminococcus torques

INTERVENTIONS:
Biological: Placebo — The placebo will consist of solely glycerol-phosphate-buffered isotonic saline.
  Arms: Placebo
Biological: Ruminococcus torques — 10^11 live bacterial cells in glycerol-phosphate-buffered isotonic saline
  Arms: Ruminococcus torques

SUMMARY:
A randomized, placebo controlled crossover study investigating the potential metabolic effects of the naturally occurring gut microbe Ruminococcus torques in healthy, overweight adults.

DETAILED DESCRIPTION:
By analyzing blood samples, indirect calorimetric as well as thermographic assessment of clavicular temperature we want to investigate whether or not the commensal gut bacterium Ruminococcus toqrues strain ATCC 27756 has any metabolic effects in healthy adults. The subjects will recieve the intervention with the live bacterium given through a duodenal feeding tube. The trial is double blinded and placebo controlled using a crossover design. Subjects will be given an intervention with either placebo or Ruminococcus on two different study days with up to six weeks of wash-out between each study day.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 40 years
* Self-reported good health
* Caucasian
* Body Mass Index > 27 kg/m^2

Exclusion Criteria:

* Any known disorder/disease that could interfere with study results or is seen as compromising to the study (as assessed by the investigator), for example diabetes, cancer or cardiovascular or kidney disease.
* Use of any daily medication as well as p.r.n. (pro re nata; not taken regularly) medication that cannot be discontinued during the trial
* Use of antibiotics during the recent three months
* Acute or chronic gastrointestinal symptoms
* Lactose intolerance
* Pregnancy - ongoing or planned
* Smoking
* Alcohol or drug abuse
* Use of creatine as dietary supplement during study period
* Plasma creatinine above the normal range (>105 μmol/L for men and >90 μmol/L for women)
* Known significant liver disease or plasma alanine transaminase concentration ≥ 3 × normal value
* Values for hemoglobin, leukocytes, or thrombocytes outside of the normal ranges

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2023-05-03 (Actual); Primary Completion 2023-09-06 (Actual); Study Completion 2023-09-14 (Actual)

PRIMARY OUTCOMES:
Matsuda Insulin Sensitivity Index | During two hours following a standard glucose solution (75g glucose in 250 ml of water) after the second dose of Ruminococcus or placebo has been given during the study day (second measurement up to six weeks later)
  Differences in calculated Matsuda Insulin Sensitivity Index between the two study days

SECONDARY OUTCOMES:
Ruminococcus Irisin-Like Peptide (RUCILP) | During the six hours of the study day (up to six weeks between study days)
  Differences in plasma RUCILP concentration between the two study days
Peptide YY | During the six hours of the study day (up to six weeks between study days)
  Differences in plasma Peptide YY concentration between the two study days
Glucose profile | During the six hours of the study day (up to six weeks between study days)
  Difference in blood glucose profile during the entirety of the study day
Resting energy expenditure | Three times during the study day for 15 minutes
  Difference in resting energy expenditure measured by indirect calorimetric
Activation of brown adipose tissue | 15 minutes 3 times during each study day
  Difference in temperature measured with thermographic camera of the collar bones
Bone dynamics | During the six hours of the study day (up to six weeks between study days)
  Differences in measures of biomarkers of bone turnover in blood
Gut microbiota | Samples taken prior to each visit (experimental days and follow-up visits)
  Changes in gut microbiota composition after each intervention
Metabolome | During the six hours of the study day (up to six weeks between study days)
  Changes is plasma metabolome after intervention
Area Under the Plasma Concentration Versus Time Curve of Gucagon-Like Peptide-1 | During the six hours of the study day (up to six weeks between study days)
  Differences in area under the curve between the two study days
Cytokine profile | During the six hours of the study day
  Differences in the cytokine profiles during the study day

OTHER OUTCOMES:
Heart rate | During the six hours of the study day (up to six weeks between study days)
  Changes in heart rate during study day
Blood pressure | During the six hours of the study day (up to six weeks between study days)
  Changes in blood pressure during study day
Various hormones related to metabolism | During the six hours of the study day (up to six weeks between study days)
  Differences in measures of various hormones during the study day
Standard hematologic blood samples | During the six hours of the study day (up to six weeks between study days) as well as one week after each study day
  Differences in measures of standard hematologic biomarkers in the blood, such as platelets
Standard clinical biochemical variables | During the six hours of the study day (up to six weeks between study days) as well as one week after each study day
  Differences in measurements of standard clinical biochemical biomarkers, such as alanine transaminase and creatinine

CONTACTS AND LOCATIONS:
Overall Officials: Oluf B Pedersen, Prof, MD, Principal Investigator — Gentofte Hospital
Locations (1):
- Gentofte Hospital, Hellerup, Denmark

IPD SHARING:
Plan to Share IPD: No